CLINICAL TRIAL: NCT00600054
Title: Phase 2 Study of Safety and Efficacy of Nimotuzumab (TheraCIM®) in Pediatric Patients With Recurrent Diffuse Intrinsic Pontine Glioma
Brief Title: Phase 2 Study of Nimotuzumab in Pediatric Recurrent Diffuse Intrinsic Pontine Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Responsible Party: Wendy Chapman, Vice President, Clinical Operations, YM BioSciences Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMB1000-013
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Recurrent Diffuse Pontine Gliomas
Keywords: Diffuse intrinsic pontine glioma; Common Terminology Criteria; Epidermal Growth factor receptor; Human antihuman antibody; pharmacokinetics; monoclonal antibody; Informed Consent Form
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental)
  Interventions: Biological: nimotuzumab (anti EGFR humanized monoclonal antibody)

INTERVENTIONS:
Biological: nimotuzumab (anti EGFR humanized monoclonal antibody) — 150 mg/m2 I.V. Induction phase: infusions once a week for 8 weeks. Consolidation phase: infusions once every 2 weeks for 10 weeks. Patients may then continue on the consolidation regimen of nimotuzumab, until disease progression or the occurrence of unacceptable toxicity.

SUMMARY:
This is a phase 2, single-arm, multi-center study, with a safety review component, designed to evaluate the efficacy and safety of nimotuzumab in approximately 44 patients with recurrent diffuse intrinsic pontine glioma (DIPG) following one previous regimen for their disease. Patients must be diagnosed with radiologically verified recurrent diffuse intrinsic pontine glioma that is measurable in at least two dimensions. Patients are eligible without histologic confirmation. Treatment regimen will consist of two phases-induction and consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients with recurrent, diffuse intrinsic pontine gliomas
* Patients should have had 2 of the following 3 neurological symptoms: cranial nerve deficit, long tract signs, ataxia and a onset prior to initial diagnosis < 6 months.
* Evidence of disease progression
* Have a Lansky or Karnofsky Performance Status of > 40
* Be between the age >3 years to < 18 years of age
* Have a tumor that is measurable radiologically
* For female patients of childbearing age: presence of a negative pregnancy test within 7 days prior to day 0.
* Use of effective contraception
* Adequate hematological, renal, and hepatic function

Exclusion Criteria:

* A history of prior use of EGFR-targeting agents (monoclonal antibodies, tyrosine kinase inhibitors)
* More than one line of treatment
* Patients with disseminated disease are not eligible
* Had radiation therapy completed within 12 weeks of enrollment
* Previous chemotherapy completed < 2 weeks prior to enrollment
* If female, is pregnant or lactating
* Has other existing serious medical conditions
* Has any condition, therapy, or medical condition, which, in the opinion of the attending physician could represent a risk for the patient or adversely affect the study objectives
* Is currently taking or planning to take other investigational drugs during the study
* Known contraindications against antibodies

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine the objective response rate | To determine response rate on week 18

SECONDARY OUTCOMES:
To evaluate the safety profile of single agent nimotuzumab in this population | safety will be evaluated after each study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bouffet, MD, Principal Investigator — The Hospital for Sick Children; Ute Bartels, MD, Principal Investigator — The Hospital for Sick Children; Sylvain Baruchel, MD, Principal Investigator — The Hospital for Sick Children
Locations (13):
- United States (10):
  - Children's Hospital/University of Colorado, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - The Sidney Kimmel Comprehensive Cancer Center, Johns Hopkins, Baltimore, Maryland
  - NYU Medical Center, Hassenfeld Clinic, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Strong Memorial Hospital, Rochester, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas/M.D. Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - The Hospital For Sick Children, Toronto, Ontario
- The Chaim Sheba Medical Center, Tel Litwinsky, Tel-Hashomer, Israel